

# STATISTICAL ANALYSIS PLAN (SAP) TEMPLATE FOR NON-INTERVENTIONAL STUDIES

# Non-Interventional Study Protocol <X9001134>

# The real world evidence on treatment patterns, effectiveness, and safety of drugs for stroke prevention in nonvalvular atrial fibrillation patients in Korea

Statistical Analysis Plan (SAP)

Version: 3.0

Author: PPD MPharm, MA, PhD PPD

Korea)

**Date**: 03-May-2018


# TABLE OF CONTENTS

| 1 | AN | MENDMENTS FROM PREVIOUS VERSION(S) | 4 |
|---|---|---|---|
| 2 | IN' | TRODUCTION | 7 |
| | 2.1<br>2.2 | STUDY DESIGNSTUDY OBJECTIVES | |
| 3 | AN | ALYSIS SETS/ POPULATIONS | 11 |
| | 3.1<br>3.2 | FULL ANALYSIS SET | |
| 4 | EN | DPOINTS AND COVARIATES | 14 |
| | 4.1<br>4.2<br>4.3<br>4.4<br>4.5 | EFFICACY/ EFFECTIVENESS ENDPOINT(S) SAFETY ENDPOINTS OTHER ENDPOINTS COVARIATES HANDLING OF MISSING VALUES | 15<br>15<br>16 |
| 5 | ST | ATISTICAL METHODOLOGY AND STATISTICAL ANALYSES | 19 |
| | 5.1<br>5.2 | STATISTICAL METHODSSTATISTICAL ANALYSES | |
| 6 | SU | MMARY OF ANALYSES | 23 |
| 7 | LIS | ST OF TABLES | 24 |
| 8 | AP | PENDIX | 25 |
| 9 | RE | FERENCES | 34 |

\_\_\_\_\_

# 1 AMENDMENTS FROM PREVIOUS VERSION(S)

| Amendment<br>number | Date | Substantial or administrative amendment | SAP section(s)<br>changed | Summary of amendment(s) | Reason | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Amendment<br>01 (V2.0) | 31Jan2018 | Substantial<br>amendment | 2.1 STUDY<br>DESIGN | Add "Comparative analyses will be performed contingent on a feasibility assessment based on the descriptive analyses." | Meet to Harmonized SAP | | | | | |
| | | | | Clarify the reference period for AF diagnosis | | | | | | |
| | | Substantial amendment | 2.2 STUDY<br>OBJECTIVES | Change phrases aligned with protocol | According to protocol amendment | | | | | |
| | | Substantial amendment | 3 ANALYSIS<br>SETS/<br>POPULATIONS | Change Inclusion & Exclusion criteria | According to protocol amendment | | | | | |
| | | Substantial amendment | 4.1 EFFICACY/<br>EFFECTIVENESS<br>ENDPOINT(S) | Add 'Hemorrhagic stroke' in operational definition | Meet to Harmonized SAP | | | | | |
| | | Substantial | 4.2 SAFETY | Change to 'Major bleeding' | Meet to Harmonized SAP | | | | | |
| | | | | | amendment | ENDPOINTS | Delete the 'Clinically relevant non-major bleeding' | | | |
| | | Substantial<br>amendment | 5.1<br>STATISTICAL<br>METHODS | Add Balance diagnostics & IPTW diagnostics | Specify the analysis method for propensity score | | | | | |
| Amendment 02 (V3.0) | 23Apr2018 | Substantial amendment | 2.Study design | Add 'other NOACs, new use of warfarin, and aspirin' | More detailed description of the objectives | | | | | |
| | | | | Delete 'aspirin-clopidogrel combination, and clopidogrel' | | | | | | |
| | | Substantial amendment | 2.2 study objectives | Delete ''to explore baseline characteristics and drug utilization patterns of antithrombotic therapies in special patients grougs (i.e., coronary intervention patients) | This secondary objective will have a separate protocol (in agreement with global HEOR team guidance) | | | | | |
| | | | | | | | | amendment codes for inclusion on ICD-10 and a KCD code is slig ICD-10 (e.g., ICD | Add ' [NOTE] KCD code is based<br>on ICD-10 and almost similar, but<br>KCD code is slightly different from<br>ICD-10 (e.g., ICD-10 is more<br>subdivided and extensive than KCD<br>code | More details on the difference<br>between ICD-10 and KCD codes<br>provided |
| | | Administrative amendment | 3. 1 Exclusion criteria | Delete ' hip or knee replacement' in<br>medical claims indicating a<br>diagnosis code of others during the<br>12-month baseline period | Conflicts with the exclusion criteria #1;duplicate | | | | | |
| | | Administrative amendment | 3. 1 Exclusion criteria | Revise #6 as 'for the comparison of "NOAC versus NOAC", and "NOAC versus warfarin, patients with any OACs (apixaban, dabigatran, rivaroxaban, or warfarin) | More clear statements for NOAC vs<br>NOAC and NOAC vs VKA<br>comparison | | | | | |

# NIS Protocol <X9001134> Statistical Analysis Plan <Version 3.0> <03 May 2018>

| Amendment<br>number | Date | Substantial or administrative amendment | SAP section(s)<br>changed | Summary of amendment(s) | Reason |
|---|---|---|---|---|---|
| | | | | in the pre-index period | |
| | | Substantial amendment | 3.1 Exclusion criteria | Revise #7 as 'for the comparison of "NOAC versus aspirin", patients with following medications in the pre-index period (from 1 year prior to the day before index date) | More clear statements for NOAC vs aspirin |
| | | Administrative amendment | 3.1 Cohorts | Add statements on dataset for<br>NOAC vs NOAC, NOAC vs<br>warfarin, NOAC vs aspirin | Details provided for each comparison cohorts |
| | | Administrative amendment | 3.1 Cohorts | Delete ' [Note] clopidogrel, aspirin,<br>clopidogrel will be included in<br>descriptive analysis' | Deleted the statement for relocation |
| | | Administrative amendment | 3.2 Subgroups | Revise as 'subgroup analysis may be considered, including but not limited to subgroup analyses by' | More broad statements to cover various topics for sub-analyses |
| | | Substantial amendment | 4.1<br>Efficacy/effectiven<br>ess endpoints | Revise to include hospitalization and CT/MRI imaging for all outcomes, more explanation on how the events were measured | Corrected errors |
| | | | | Add 'individual outcome of primary outcome' Deleted myocardial infarction | |
| | | Substantial amendment | 4.2 Safety endpoints | Add statement regarding main subdiagnosis codes being used Add 'hospitalization and brain | More clear statements added |
| | | | | CT/MRI to identify ICH' Add individual outcome of major bleeding, clinical events preceding each pattern, compliance | |
| | | Administrative amendment | 5.1 Descriptive analysis | Add 'the proportion of antithrombotics at index date will be examined' | More details on the treatment pattern provided |
| | | Administrative amendment | 5.1 Multivariate analysis | Specific comparison cohorts for analysis | More clear statements included |
| | | | | Add statements on covariate adjustment propensity score | |
| | | | | Delete references used under IPTW diagnostics | |
| | | | | Add statements for each comparison cohorts | |
| | | | 5.1 Statistical methods | Additional sensitivity analysis | Perform IPTW using the propensity score derived from multinomial model |
| | | Substantial amendment | 5.2 Statistical analyses | Add ' other propensity score method will also be used' | More clear statements included |


# NIS Protocol <X9001134> Statistical Analysis Plan <Version 3.0> <03 May 2018>

| Amendment<br>number | Date | Substantial or administrative amendment | SAP section(s)<br>changed | Summary of amendment(s) | Reason |
|---|---|---|---|---|---|
| | | Administrative amendment | 6.Summary of analyses | Delete 'myocardial infarction' | Removed for accuracy |
| | | Administrative amendment | 8. Appendix | Add statements regarding bleeding outcomes and procedures codes | More details provided |
| | | Substantial amendment | Appendix 2. Data derivation details | Revise codes for effectiveness and safety outcomes codes | Input codes according to changes in the outcome endpoints |
| | | Substantial amendment | Table 13.<br>Exclusion criteria | Add codes for each conditions | More details provided |
| | | Substantial amendment | Table 14. Blood transfusion codes | Add codes for Korean procedure codes used | More details provided |

\_\_\_\_\_\_

#### 2 INTRODUCTION

Atrial fibrillation (AF) is the most common persistent arrhythmia, and its prevalence has been estimated to be 1-2% of the general population, with a progressive increase (1). AF increases the risk of ischemic stroke by five-fold and is associated with 15% of stroke for all age groups and 30% in patients aged 80 years and older (2). Patients with AF-related ischemic stroke have higher recurrent risk, morbidity, and mortality as compared to patients with other types of stroke (3). Thus, current clinical guidelines for AF emphasize stroke prevention in patients with AF, in the presence of stroke risk factors (4). Effective stroke prevention essentially requires oral anticoagulants (OAC) therapy. Vitamin K antagonists (i.e., warfarin) effectively decrease the risk for thromboembolic events in patients with AF (5). However, vitamin K antagonists have several limitations, including need for regular blood monitoring and possibility for food or drug interactions. This had led to the quest for new OACs that would be more safe and effective than warfarin (6). In randomized controlled trials, NOACs demonstrated noninferior or superior reduction in stroke and systemic embolism when compared to warfarin (7-10).

Physicians now have a choice between the available NOACs but have relatively little evidence to guide their decision-making because of no head-to-head trials of these drugs. In addition, there have been far fewer studies on efficacy and safety outcomes of NOACs. The nationwide claims database in Korea can provide an opportunity to study comparative effectiveness and safety outcomes of NOACs in patients with atrial fibrillation in Korea.

# 2.1 STUDY DESIGN

This study will use a retrospective cohort design in which the treatment effectiveness and safety outcomes of new use of NOACs compared to other NOACs, new use of warfarin, and aspirin will be estimated in patients with atrial fibrillation using the Korean Health Insurance Review & Assessment Service (HIRA) database. Comparative analyses will be performed contingent on a feasibility assessment based on the descriptive analyses. Propensity score method and Cox proportional hazards models will be used to account for selection bias, differences in follow-up time, and right data censoring. This will allow us to minimize selection bias and confounding bias and provide outcome data amenable to rapid clinical interpretation (i.e., time-to-event analysis, hazard ratios). Furthermore, HIRA database will allow us to preserve the population-based longitudinal data collection advantages. The overall study design is described in Figure 1.



Figure 1. Study design scheme

# Study population

Subjects with atrial fibrillation (between January 1, 2007 up to and including the index date\*) who newly initiated NOACs, warfarin, or used aspirin between July 1, 2015 and November 30, 2016 in the Korean Health Insurance Review & Assessment Service (HIRA) database.

\*Index date is the first prescription date of study drugs, including NOACs, warfarin, and aspirin.

#### Data source

South Korea has a universal health coverage system that the National Health Insurance covers approximately 97% of the overall South Korean population. The claims data of Health Insurance Review & Assessment Service (HIRA) contains 46 million patients per year that account for 90% of the total population in Korea and include claims from almost 80,000 healthcare service providers across South Korea as of 2011.

The claims data of HIRA includes patients' diagnosis, treatment, procedures, surgical history, and prescription drugs which provide a valuable resource for healthcare service research. Data elements captured in the HIRA database include patient-level demographic and plan enrollment information (e.g., start and stop dates of health plan enrollment), date-stamped (month and year) inpatient and outpatient medical claims (e.g., diagnosis codes, procedure codes, provider specialty), and pharmacy claims (e.g., prescription fill/refill dates, drug name/code, dosage). While procedure codes that identify patient receipt of laboratory tests are available, actual laboratory values and test results are not available.

The HIRA database has unique attributes that make it a useful data source for this study. The key advantage of the HIRA database relative to other potential data sources (e.g., medical chart review) is that it is a population level data including most of Korean population and it will provide a large analytic sample and provide accurate claim-level treatments pattern and health care utilization across all provider settings (e.g., inpatient, outpatient, pharmacy) in patients' spectrum of care.

One key limitation of the HIRA database is that it does not include clinical variables such as laboratory values and clinical markers. To overcome this limitation, the Charlson comorbidity index and overall healthcare utilization observed during the pre-index period will be used as proxy measures to incorporate the overall health status of the individual patients.

\_\_\_\_\_

#### 2.2 STUDY OBJECTIVES

# Primary objectives

- 1. To explore baseline characteristics and drug utilization patterns in patients with nonvalvular atrial fibrillation (NVAF) who newly initiated NOACs, warfarin, or used aspirin
  - Demographic and clinical characteristics: Age, sex, types of health insurance, CHA<sub>2</sub>DS<sub>2</sub>-VASc score, HAS-BLED score, Charlson Comorbidity Index score, etc.
  - Descriptions of index treatment: Types of medication received, index dose intensity
  - o Drug utilization pattern: Each patient will be followed-up until the first treatment modification occurs, or study ends (November 30, 2016).
- 2. To compare effectiveness including hemorrhagic stroke, ischemic stroke and systemic embolism of antithrombotic therapies in patients with NVAF with the following antithrombotic therapies: NOACs, warfarin, and aspirin
  - Primary effectiveness outcome: Composite of hemorrhagic stroke, ischemic stroke, and systemic embolism
  - Secondary effectiveness outcomes: Individual outcome of hemorrhagic stroke, ischemic stroke, and systemic embolism
- 3. To compare safety of anti-thrombotic therapies in patients with NVAF with the following antithrombotic therapies: NOACs, warfarin, and aspirin
  - o Primary safety outcome: Major bleeding including gastrointestinal bleeding or intracranial bleeding and other bleeding
  - Secondary safety outcomes: Individual outcome of major bleeding

[NOTE] comparative analyses will be performed contingent on a feasibility assessment based on the descriptive analyses.

# Secondary objectives

- 1. To explore and understand more detailed drug utilization patterns
  - Standard dose versus reduced dose

- o Pattern of usage (i.e., switching, discontinuation) and clinical events preceding the pattern
- o Compliance (i.e., medication possession ratio)
- 2. To compare effectiveness and safety of antithrombotic therapies versus not using therapies among low risk patients (low score of CHA<sub>2</sub>DS<sub>2</sub>-VASc)

# 3 ANALYSIS SETS/ POPULATIONS

# 3.1 FULL ANALYSIS SET

#### Inclusion criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

- 1. Patients aged 18 years or older on the index date
- 2. Patients had ≥1 medical claim for AF (refer to Table 1) before or on the index date with at least one hospitalization or at least two outpatient visits:

# [Diagnosis codes for inclusion criteria]

| KCD-6 <sup>1)</sup> | KCD-7 <sup>2)</sup> |
|---|---|
| I48 (Atrial fibrillation and flutter) | I48 (Atrial fibrillation and flutter) |
| I480 (Atrial fibrillation) | I480 (Paroxysmal atrial fibrillation) |
| I481 (Atrial flutter) | I481 (Persistent atrial fibrillation) |
| | I482 (Chronic atrial fibrillation) |
| | I483 (Typical atrial flutter) |
| | I484 (Atypical atrial flutter) |
| | I489 (Atrial fibrillation and atrial flutter, |
| | unspecified) |

KCD-6, Korean version of ICD-10 (6<sup>th</sup> revision); KCD-7, Korean version of ICD-10 (7<sup>th</sup> revision)

- 1) KCD-6 diagnosis codes will be used from 1 July 2015 to 31 December 2015.
- 2) KCD-7 diagnosis codes will be used from 1 January 2016 to 30 November 2016.

[NOTE] KCD code is based on ICD-10 and almost similar, but KCD code is slightly different from ICD-10 (e.g., ICD-10 is more subdivided and extensive than KCD code).

3. Patients prescribed aspirin, warfarin, or NOACs in intake period (from July 1, 2015 to November 30, 2016)

[Note] NOACs include apixaban, dabigatran and rivaroxaban.

# Exclusion criteria

Patients meeting any of the following criteria will not be included in the study.

- 1. Medical claims indicating diagnosis or procedure for hip/knee replacement surgery within 6 weeks prior to index date
- 2. Medical claims indicating a diagnosis code indicative of rheumatic mitral valvular heart disease, mitral valve stenosis during the 12-month baseline period
  - (Valvular AF / Prosthetic heart valves)
- 3. Medical claims indicating a diagnosis code of VTE (Venous thromboembolism) during the 12-month baseline period
- 4. Medical claims indicating a diagnosis or procedure code of transient AF, or cardiac surgery during the 12-month baseline period
  - (Thyrotoxicosis, Hypertrophic cardiomyopathy, elective defibrillation, radiofrequency ablation, or left atrial appendage occlusion)
- 5. Medical claims indicating a diagnosis code of others during the 12-month baseline period
  - (End-stage chronic kidney disease / Kidney transplant / Dialysis / Pericarditis)
- 6. For the comparison of "NOAC versus NOAC", and "NOAC versus warfarin", patients with any OACs (apixaban, dabigatran, rivaroxaban, or warfarin) in the pre-index period (from 1 year prior to the day before index date)
  - o [NOTE] Patients prescribed antiplatelets in the pre-index period will not be excluded.
- 7. For the comparison of "NOAC versus aspirin", patients with following medications in the pre-index period (from 1 year prior to the day before index date)
  - o NOAC user: OACs (apixaban, dabigatran, rivaroxaban, warfarin)
  - o Aspirin user: none
  - o [NOTE] NOAC user is defined as OAC naïve user and aspirin user is allowed to have OACs or antiplatelets in the pre-index period.

# **Cohorts**

To avoid increasing type I error when multiple comparisons occur, this full analysis set will be splitted into multiple sub-analysis sets as follows:

- 1. NOAC vs NOAC (both as OAC naïve users)
  - A. Sub-dataset 1: patients with index treatment of apixaban and patients with index treatment of dabigatran
  - B. Sub-dataset 2: patients with index treatment of apixaban and patients with index treatment of rivaroxaban
  - C. Sub-dataset 3: patients with index treatment of dabigatran and patients with index treatment of rivaroxaban

[NOTE] The index date will be defined as date of the first prescription of NOAC in patients with NVAF. To identify new users, a look-back observation period from 1 year prior to the day before the index date will be used and must indicate no OAC use during this period. The diagnosis date of NVAF could occur from January 1, 2007 up to and including the index date.

- 2. NOAC vs warfarin (both as OAC naïve users)
  - A. Sub-dataset 4: patients with index treatment of apixaban and patients with index treatment of warfarin
  - B. Sub-dataset 5: patients with index treatment of dabigatran and patients with index treatment of warfarin
  - C. Sub-dataset 6: patients with index treatment of rivaroxaban and patients with index treatment of warfarin

[NOTE] The index date will be defined as date of the first prescription of NOAC or warfarin in patients with NVAF. To identify new users, a look-back observation period from 1 year prior to the day before the index date will be used and must indicate no OAC use during this period. The diagnosis date of NVAF could occur from January 1, 2007 up to and including the index date.

- 3. NOAC (OAC naïve user) vs aspirin (no restrictions of antiplatelet or OAC use in the pre-index period)
  - A. Sub-dataset 7: patients with index treatment of apixaban and patients with index treatment of aspirin
  - B. Sub-dataset 8: patients with index treatment of dabigatran and patients with index treatment of aspirin
  - C. Sub-dataset 9: patients with index treatment of rivaroxaban and patients with index treatment of aspirin

\_\_\_\_\_

[NOTE] The index date will be defined as date of the first prescription of NOAC or aspirin in patients with NVAF during the intake period (from July 1, 2015 to November 30, 2016). To identify NOAC users, a look-back observation period from 1 year prior to the day before the index date will be used and must indicate no OAC use during this period. However, OAC use or antiplatelet use during a look-back observation period from 1 year prior to the day before the index date will be allowed for aspirin users. The diagnosis date of NVAF could occur from January 1, 2007 up to and including the index date.

Each patient was followed until discontinuation or switching of index treatment, outcome occurrence, or study ends (November 30, 2016).

# 3.2 SUBGROUPS

Subgroup analysis may be considered, including but not limited to subgroup analyses by CHA<sub>2</sub>DS<sub>2</sub>-VASc score, HAS-BLED score and the dose of index treatment.

# 4 ENDPOINTS AND COVARIATES

# 4.1 EFFICACY/ EFFECTIVENESS ENDPOINT(S)

**Table 1. Effectiveness Endpoints** 

| Variable | Role | Operational definition |
|---|---|---|
| Stroke/Systemic embolism | Primary effectiveness<br>outcome | Hemorrhagic stroke, ischemic stroke and systemic embolism requiring hospitalization will be identified using hospital claims which had a hemorrhagic stroke, ischemic stroke or systemic embolism code whichever came first (i.e., the first occurred event will be used). All KCD diagnosis codes (main and sub-diagnosis codes) will be used. Especially, hospitalization and brain CT or MRI codes will be needed to identify ischemic stroke and hemorrhagic stroke. For systemic embolism, hospitalization and any CT or MRI codes will be used (Appendix 2, Table 7). |
| Individual outcome of primary outcome | Secondary effectiveness outcome | Individual outcome of hemorrhagic stroke (diagnosis codes in all main and sub-diagnosis codes + hospitalization + brain CT or MRI), ischemic stroke (diagnosis codes in all main and sub-diagnosis codes + hospitalization + brain CT or MRI), and systemic embolism (diagnosis codes |


| Variable | Role | Operational definition |
|---|---|---|
| | | in all main and sub-diagnosis codes +<br>hospitalization + any CT or MRI) |

# 4.2 SAFETY ENDPOINTS

**Table 2. Safety Endpoints** 

| Variable | Role | Operational definition |
|---|---|---|
| Major bleeding | Primary safety outcome | Bleeding requiring hospitalization will be identified using hospital claims which had a bleeding diagnosis code as the first occurred KCD code and it will be consisted of intracranial hemorrhage (ICH) and gastrointestinal (GI) bleeding, and other bleeding (Appendix 2, Table 8). All KCD diagnosis codes (main and subdiagnosis codes) will be used. Especially, hospitalization and brain CT or MRI codes will be needed to identify ICH. |
| Individual outcome of major bleeding | Secondary safety outcome | Individual outcome of ICH (diagnosis codes in all main and sub-diagnosis codes + hospitalization + brain CT or MRI), gastrointestinal bleeding (diagnosis codes in all main and sub-diagnosis codes + hospitalization), and other bleeding (diagnosis codes in all main and sub-diagnosis codes + hospitalization) |

# 4.3 OTHER ENDPOINTS

**Table 3. Other Endpoints** 

| Variable | Role | Operational definition |
|---|---|---|
| Discontinuation | Outcome | Discontinuation is defined as the first day of a period of at least 30 consecutive days after the calculated time to finishing the pack based on pack size and number of tablets per day. The date of discontinuation will be the end date of the last filled prescription before the treatment gap. |
| Switching | Outcome | A switch among anticoagulants will be defined as a prescription filled for non-index OAC within 30 |

| Variable | Role | Operational definition |
|---|---|---|
| | | days after the date of discontinuation. |
| Clinical events preceding each pattern | Outcome | Types of event* preceding each pattern (i.e., discontinuation, switching) [*Note] Events will include but not limited to (1) serious clinical events where physicians might consider changing anticoagulants (e.g., thromboembolic events (e.g., stroke/systemic embolism, venous thromboembolism [codes in Table 7]), major bleeding [codes in Table 8]); (2) the occurrence of a contraindication for OACs (e.g., valvular atrial fibrillation, severe kidney disease); and (3) procedure for atrial fibrillation that might not require OACs (e.g., elective defibrillation, radiofrequency ablation, and left atrial appendage occlusion [codes in Table 13]). |
| Compliance (medication possession ratio, MPR) | Outcome | Medication possession ratio (MPR) will be calculated as total days of index treatment dispensed / 365 days of study follow-up. Patients with an MPR greater than 1 will be capped at 1. |

# 4.4 COVARIATES

**Table 4. Baseline Variables** 

| Variable | Role | Operational definition |
|---|---|---|
| Age | Baseline<br>characteristic<br>and potential<br>confounder | Age at index date |
| Sex | Baseline<br>characteristic<br>and potential<br>confounder | 1. Male 2. Female |
| Types of health insurance | Baseline<br>characteristic<br>and potential<br>confounder | Types of health insurance divided as the following: 1. National Health Insurance 2. Medical aid |

| Variable | Role | Operational definition |
|---|---|---|
| $\mathrm{CHA}_2\mathrm{DS}_2	ext{-VASc}$ | Baseline<br>characteristic<br>and potential<br>confounder | CHA <sub>2</sub> DS <sub>2</sub> -VASc as continuous data or dichotomous data. The score will be calculated using the following KCD codes (Appendix 2, Table 9): 1. Congestive heart failure 2. Hypertension 3. Diabetes mellitus 4. Stroke/TIA/TE 5. Vascular disease 6. Age ≥ 75 7. Age 65-74 8. Female |
| HAS-BLED | Baseline<br>characteristic<br>and potential<br>confounder | HAS-BLED as continuous data or dichotomous data. The score will be calculated using the following KCD codes (Appendix 2, Table 10): 1. Hypertension 2. Abnormal renal function 3. Abnormal liver function 4. Stroke 5. Bleeding history or predisposition: refers to any bleeding codes 6. Age > 65 7. Antiplatelet or NSAID use 8. Alcoholism [Note] Labile international normalized ratio is not available in HIRA data and does not apply to patients on aspirin, or NOACs, so the modified HAS-BLED score has a maximum value of 8 instead of 9. |
| Charlson Comorbidity Index | Baseline<br>characteristic<br>and potential<br>confounder | Charlson Comorbidity Index as continuous data or dichotomous data. The index will be calculated using the following KCD codes (Appendix 2, Table 11): |

| Variable | Role | Operational definition |
|---|---|---|
| | | Myocardial infarction |
| | | 2. Congestive heart failure |
| | | 3. Peripheral vascular disease |
| | | 4. Cerebrovascular disease |
| | | 5. Dementia |
| | | 6. Chronic pulmonary disease |
| | | 7. Rheumatic disease |
| | | 8. Peptic ulcer disease |
| | | 9. Mild liver disease |
| | | 10. Diabetes without chronic complication |
| | | 11. Diabetes with chronic complication |
| | | 12. Hemiplegia or paraplegia |
| | | 13. Renal disease |
| | | Any malignancy, including lymphoma and leukemia, except malignant neoplasm of skin |
| | | 15. Moderate or severe liver disease |
| | | 16. Metastatic solid tumor |
| | | 17. AIDS/HIV |
| | | It will be consisted of the following (Appendix 2, Table 12): |
| | | 1. NSAIDs |
| Baseline Medication Use | Baseline characteristic and potential | 2. Antiplatelet |
| | | 3. PPI |
| | confounder | 4. H <sub>2</sub> -receptor antagonists |
| | | 5. Antiarrhythmics |
| | | 6. Digoxin |

| Variable | Role | Operational definition |
|----------|------|------------------------|
| | | 7. Statins |

#### 4.5 HANDLING OF MISSING VALUES

After examining the characteristics of missing values, we will determine whether we can remove observations with missing values from the dataset. Basically, subjects with missing values of covariates will not contribute to the analysis.

# 5 STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES

#### 5.1 STATISTICAL METHODS

# **Descriptive Analysis:**

- O All outcome variables will be summarized descriptively through the tabular and graphical display of mean values, medians, ranges, and standard deviations for continuous variables of interest and frequency distributions for categorical variables.
- O The proportion of antithrombotics (aspirin, clopidogrel, aspirin and clopidogrel combination, warfarin, NOACs) at index date will be examined.
- O Appropriate tests (e.g., t-test, chi-square test) will be used based on the distribution of the measure. The p < 0.05 considered significant.

# **Multivariate Analysis:**

# Propensity score method

The estimation of propensity score will be performed to control for confounders in each sub-dataset: (1) each NOAC versus NOAC; (2) each NOAC versus warfarin; (3) each NOAC versus aspirin.

Propensity scores are estimated by logistic regression analyses that incorporate potential treatment predictors as independent variables and types of index treatment as dependent variable (e.g., apixaban=1, warfarin=0). Covariates in the logistic regression model will

include variables such as age, sex, CCI score, CHA<sub>2</sub>DS<sub>2</sub>-VASc score, HAS-BLED score, and comorbidities, but the final list of these covariates will be discussed and determined after reviewing the results of descriptive analysis of the pre-matched datasets. Further, we will report the *c*-statistic of the propensity score that indicates the degree to which the propensity score model discriminates between treated patients and untreated patients.

After estimation of propensity score, we will perform propensity score matching (PSM). 1:1 matching without replacement will be performed.

The populations would be first matched using PSM according to their index treatment. For these matched populations we should then explore the proposed subgroups by: making an assessment of patient numbers in the subgroups and checking that patient characteristics are still similar between the index treatments in the subgroups. If they are similar, then conduct interaction term analysis is being conducted to determine whether the treatment effect varies between the subgroups. If the populations are no longer similar in characteristics, then re-matching via PSM will be performed for the subgroups.

Covariate adjustment using propensity score will also be performed. This approach has an advantage of using the whole observations whereas matching approach uses part of observations which were successfully matched.

# Inverse probability of treatment weighted (IPTW)

We will perform an inverse probability of treatment weighted (IPTW) analysis. Every person will be weighted by the inverse of the probability of receiving the treatment actually received (i.e., PS in the treated and (1-PS) in the untreated).

# Balance diagnostics

We will compare and assess the balance of baseline variables (e.g., continuous variable, dichotomous variable, interaction terms, or squares of continuous variable) between treated and control subjects in the weighted sample using standardized difference (Austin et al., 2015).

# IPTW diagnostics

The distribution of weights will be carefully checked because some patients, those treated contrary to prediction, may receive very large weights (11, 12). To address the presence of extreme weights, we will consider several approaches, including use of stabilized weights, or trimmed or truncated weights (11-13). The stabilized weights will be implemented based on the following equation (11):

# IPTW stabilized=E\*PE/PS + (1-E)\*(1-PE)/(1-PS)

- E: treatment (E=1), no treatment (E=0).
- PE: overall marginal prevalence of the treatment exposure.
- PS: estimated propensity score.

Balances between treatment groups will be evaluated by the standardized differences of all covariates, using a threshold of 0.1 to determine an imbalance.

# Cox proportional hazards model

Cox proportional hazards model will be used to compare event rates between the treatment groups, with warfarin or antiplatelets as the primary reference in each subdataset: (1) each NOAC versus NOAC; (2) each NOAC versus warfarin; (3) each NOAC versus aspirin.

Cox model stratification (dummy variable method and true stratification method) will be performed to examine whether the stratum-to-stratum differences exist. To check the proportional hazards assumption, we will employ both the graphical methods (i.e., loglog plot, observed-expected plot, Schoenfeld residual plot) and statistical tests using the time-dependent covariate. If the assumption does not meet, we will employ either a stratified model or an interaction term between time and variable of interest (i.e., treatment indicator).

The variables included in the model will be finalized after attempting model building process. Potential interactions will also be considered.

The hazard ratio and 95% confidence interval will be provided.

# **Sensitivity Analysis**

Sensitivity analysis of performing IPTW using the propensity score derived from multinomial model will be conducted.

# 5.2 STATISTICAL ANALYSES

O Patients with aspirin, warfarin, and NOACs will be matched via propensity-score method. Patients will be matched on patient demographics (i.e., age, sex) and clinical (i.e., CHA<sub>2</sub>DS<sub>2</sub>-VASc score, Charlson Comorbidity Index score, etc.) variables. Other propensity score method (i.e., covariate adjustment, IPTW) will


also be used. Standardized difference will be used to assess the balance of variables after matching. A standardized difference < 10% will be considered acceptable.

• A Cox proportional hazards model, to account for differences in follow-up time and right data censoring, will be used to compare effectiveness and safety outcomes between treatment groups.

# 6 SUMMARY OF ANALYSES

| Outcome | Supports Protocol Objective<br>Number | Statistical Method | Covariates/ Strata |
|---|---|---|---|
| Baseline characteristics and drug utilization patterns | 1 | Chi-square test, t-test | Demographic and clinical characteristics, including baseline comorbidities |
| Stroke/systemic embolism | 2 | Propensity score method,<br>Cox proportional hazards model | Demographic and clinical characteristics, including baseline comorbidities |
| Major bleeding | 3 | Propensity score method,<br>Cox proportional hazards model | Demographic and clinical<br>characteristics, including baseline<br>comorbidities |

# 7 LIST OF TABLES

| Table 1. Effectiveness Endpoints | 14 |
|-------------------------------------------------------|----|
| Table 2. Safety Endpoints | 15 |
| Table 3. Other Endpoints | |
| Table 4. Baseline Variables | |
| Table 5. Baseline characteristics (example) | 25 |
| Table 6. Hazard ratios for each comparison (example) | 26 |
| Table 7. Effectiveness Outcomes Codes | |
| Table 8. Safety Outcomes Codes | 28 |
| Table 9. CHA <sub>2</sub> DS <sub>2</sub> -VASc Score | |
| Table 10. HAS-BLED Score | 29 |
| Table 11. Charlson Comorbidity Index | 30 |
| Table 12. Baseline Medications | 31 |
| Table 13. Exclusion Criteria | 31 |
| Table 14. Blood Transfusion Codes | 32 |

\_\_\_\_\_

# 8 APPENDIX

# 8.1 APPENDIX 1. TABLE SHELLS

Table 5. Baseline characteristics (example)

| | Apixaban | Warfarin |
|----------------------------------------------|----------|-----------|
| | (n=XX) | (n=XX) |
| Age – mean, SD | | |
| Gender | | |
| Female | | |
| Male | | |
| Insurance type | | |
| National Health | | |
| Insurance | | |
| Medical Aid | | |
| CHA <sub>2</sub> DS <sub>2</sub> -VASc score | | |
| Mean (SD) | | |
| 0-1 | | |
| 2 | | |
| 3 | | |
| 4 | | |
| ≥5 | | |
| HAS-BLED | | |
| Mean (SD) | | |
| 0-2 | | |
| ≥3 | | |
| Charlson Comorbidity | | |
| Index | | |
| Mean (SD) | | |
| 0-1 | | |
| 2-3 | | |
| ≥4 | | |
| Comorbidities | | |
| Stroke/TIA | | |
| Systemic embolism | | |
| MI | | |
| Bleeding* | | |
| Hypertension | | |
| Diabetes mellitus | | |
| CAD | | |
| | 1 | D 25 -624 |


| | Apixaban (n=XX) | Warfarin<br>(n=XX) |
|------------------------|-----------------|--------------------|
| PAD | , | |
| Heart failure | | |
| COPD | | |
| Renal disease | | |
| Medication use | | |
| NSAIDs | | |
| Antiplatelet | | |
| PPI | | |
| H2-receptor antagonist | | |
| Digoxin | | |
| Statin | | |
| Antiarrhythmics | | |

<sup>\*</sup>Bleeding will be identified as the same with the definition of major bleeding outcomes and the transfusion procedure codes (see Table 14 for codes).

Table 6. Hazard ratios for each comparison (example)

| | Apixaban<br>(n=XX) | Warfarin<br>(n=XX) | Apixaban vs warfarin (n=XX) | |
|---|---|---|---|---|
| | Event rate | Event rate | HR (95% CI) | P value |
| Effectiveness endpoints | | | | |
| Stroke/systemic embolism | | | | |
| Safety endpoints | | | | |
| Major bleeding | | | | |

# APPENDIX 2. DATA DERIVATION DETAILS

**Table 7. Effectiveness Outcomes Codes** 

| Type | KCD Code or Procedure Code |
|---|---|
| Hemorrhagic stroke* | I60, I61, I62, I690, I691, I692 |
| Ischemic stroke* | G459, I63, I693 |
| Systemic embolism** | 174 |
| *Brain CT/MRI | CT: HA441, HA451, HA461, HA471, HA851 |
| | MRI: HE101, HE102, HE135, HE201, HE202, HE235, HE301, HE302, HE401, HE402, HE501, HE502, HE535 |
| **Any CT/MRI | HE301, HE302, HE401, HE402, HE501, HE502, HE535 CT: HA401, HA402, HA403, HA404, HA405, HA406, HA407, HA408, HA409, HA410, HA411, HA412, HA413, HA414, HA415, HA416, HA424, HA425, HA434, HA435, HA443, HA443, HA445, HA446, HA445, HA446, HA447, HA448, HA449, HA453, HA456, HA457, HA458, HA459, HA463, HA464, HA465, HA466, HA467, HA468, HA469, HA473, HA474, HA475, HA476, HA477, HA478, HA479, HA496, HA497, HA801, HA805, HA809, HA813, HA834, HA835, HA853, HA856, HA857, HA858, HA859, S4852 MRI: HE103, HE104, HE105, HE106, HE107, HE108, HE109, HE110, HE111, HE112, HE113, HE114, HE115, HE116, HE117, HE118, HE119, HE120, HE121, HE122, HE123, HE124, HE125, HE126, HE127, HE128, HE129, HE130, HE131, HE132, HE133, HE134, HE136, HE137, HE138, HE139, HE140, HE141, HE142, HE203, HE204, HE205, HE206, HE207, HE208, HE209, HE210, HE211, HE212, HE213, HE214, HE215, HE216, HE217, HE218, HE219, HE220, HE221, HE222, HE223, HE224, HE225, HE226, HE227, HE228, HE229, HE230, HE231, HE232, HE233, HE234, HE236, HE237, HE238, HE239, HE240, HE241, HE303, HE304, HE305, HE306, HE307, HE308, HE309, HE310, HE311, HE312, HE313, HE314, HE315, HE316, HE317, HE318, HE319, HE320, HE321, HE322, HE323, HE324, HE325, HE326, HE327, HE328, HE329, HE330, HE311, HE312, HE313, HE314, HE315, HE316, HE317, HE318, HE319, HE320, HE321, HE322, HE323, HE324, HE325, HE326, HE327, HE328, HE329, HE330, HE311, HE312, HE313, HE314, HE315, HE316, HE317, HE318, HE319, HE320, HE321, HE322, HE323, HE324, HE325, HE326, HE327, HE328, HE329, HE330, HE331, HE314, HE315, HE313, HE314, HE315, HE333, HE334, HE324, HE325, HE326, HE327, HE328, HE329, HE330, HE331, HE332, HE333, HE334, HE403, HE404, HE330, HE331, HE332, HE333, HE334, HE403, HE404, HE330, HE331, HE332, HE333, HE334, HE403, HE404, |
| | HE405 ,HE406, HE407, HE408, HE409, HE410, HE411, HE412, HE413, HE414, HE415, HE416, HE417, HE418, |


| HE419, HE420, HE421, HE422, HE423, HE424, HE425, |
|--------------------------------------------------|
| HE426, HE427, HE428, HE429, HE430, HE431, HE432, |
| HE433, HE434, HE503, HE504, HE505, HE506, HE507, |
| HE508, HE509, HE510, HE511, HE512, HE513, HE514, |
| HE515, HE516, HE517, HE518, HE519, HE520, HE521, |
| HE522, HE523, HE524, HE525, HE526, HE527, HE528, |
| HE529, HE530, HE531, HE532, HE533, HE534, HE536, |
| HE537, HE538, HE539, HE540, HE541, HF101, HF102, |
| HF104, HF105, HF106, HF107, HF201, HF202, HF305, |
| HF306 |

<sup>\*</sup>Brain CT/MRI will be used to define hemorrhagic stroke and ischemic stroke.

**Table 8. Safety Outcomes Codes** 

| Туре | KCD Code or Procedure Code |
|---|---|
| Intracranial | I60, I61, I62, I690, I691, I692, S064, S065, S066, S068 |
| haemorrhage* | |
| Gastrointestinal bleeding | I850, I983, K2211, K226, K228, K250, K252, K254, K256, |
| | K260, K262, K264, K266, K270, K272, K274, K276, K280, |
| | K282, K284, K286, K290, K3181, K5521, K625, K920, |
| | K921, K922 |
| Other bleeding | D62, H448, H3572, H356, H313, H210, H113, H052, H470, |
| | H431, I312, N020-N029, N421, N831, N857, N920, N923, |
| | N930, N938, N939, M250, R233, R040, R041, R042, R048, |
| | R049, T792, T810, N950, R310, R311, R318, R58, T455, |
| | Y442, D683 |
| *Brain CT/MRI | CT: HA441, HA451, HA461, HA471, HA851 |
| | MRI: HE101, HE102, HE135, HE201, HE202, HE235, |
| | HE301, HE302, HE401, HE402, HE501, HE502, HE535 |

<sup>\*</sup>Brain CT/MRI will be used to define intracranial hemorrhage.

<sup>\*\*</sup>Any CT/MRI will be used to define systemic embolism.

Table 9. CHA<sub>2</sub>DS<sub>2</sub>-VASc Score

| Condition | KCD code | Point |
|--------------------------|--------------------|-------|
| Congestive heart failure | 150 | 1 |
| Hypertension | I10-I15 | 1 |
| Age | 75+ years | 2 |
| Diabetes | E10-E14 | 1 |
| Stroke | I63, I693 G459 | 2 |
| Vascular disease | I21, I252, I70-I73 | 1 |
| Age | 65-74 years | 1 |
| Sex | Female | 1 |

# **Table 10. HAS-BLED Score**

| Condition | KCD code | Point |
|---|---|---|
| Hypertension | I10-I15 | 1 |
| Abnormal renal function | N183, N184 | 1 |
| Abnormal liver function | B15-B19, C22, D684, I982, I983, K70-K77, Z944 | 1 |
| Stroke | I63, I693, G459 | 1 |
| Bleeding history or Predisposition* | Codes in Table 8 | 1 |
| Labile INR | Not measurable | Not applicable |
| Elderly | 65+ years | 1 |
| Drug therapy | Antiplatelets, NSAIDs | 1 |
| Alcoholism | E244, F10, G312, G621, G721, I426, K292,<br>K70, K860, O354, P043, Q860, T510, X45,<br>X65, Y15, Y90-Y91, Z502, Z714, Z721 | 1 |

<sup>\*</sup> Blood transfusion will also be used to define other bleeding history (see Table 14 for blood transfusion codes).

\_\_\_\_\_\_

**Table 11. Charlson Comorbidity Index** 

| Condition | KCD code | Point |
|---|---|---|
| Cerebrovascular disease | G45.x, G46.x, H34.0, I60.x-I69.x | 1 |
| Congestive heart failure | I09.9, I11.0, I13.0, I13.2, I25.5, I42.0, I42.5-<br>I42.9, I43.x, I50.x, P29.0 | 1 |
| Chronic pulmonary disease | I27.8, I27.9, J40.x–J47.x, J60.x–J67.x, J68.4, J70.1, J70.3 | 1 |
| Dementia | F00.x–F03.x, F05.1, G30.x, G31.1 | 1 |
| Diabetes without chronic complication | E10.0, E10.1, E10.6, E10.8, E10.9, E11.0,<br>E11.1, E11.6, E11.8, E11.9, E12.0, E12.1,<br>E12.6, E12.8, E12.9, E13.0, E13.1, E13.6,<br>E13.8, E13.9, E14.0, E14.1, E14.6, E14.8,<br>E14.9 | 1 |
| Mild liver disease | B18.x, K70.0-K70.3, K70.9, K71.3-K71.5, K71.7, K73.x, K74.x, K76.0, K76.2-K76.4, K76.8, K76.9, Z94.4 | 1 |
| Myocardial infection | I21.x, I22.x, I25.2 | 1 |
| Peripheral vascular disease | I70.x, I71.x, I73.1, I73.8, I73.9, I77.1, I79.0, I79.2, K55.1, K55.8, K55.9, Z95.8, Z95.9 | 1 |
| Peptic ulcer disease | K25.x–K28.x, | 1 |
| Rheumatologic disease | M05.x, M06.x, M32.x–M34.x M31.5M35.1, M35.3, M36.0 | 1 |
| Diabetes with chronic complication | E10.2–E10.5, E10.7, E11.2–E11.5, E11.7, E12.2-E12.5, E12.7, E13.2–E13.5, E13.7, E14.2–E14.5, E14.7 | 2 |
| Hemiplegia or paraplegia | G04.1, G11.4, G80.1, G80.2, G81.x, G82.x, G83.0-G83.4, G83.9 | 2 |
| Any malignancy, including leukemia and lymphoma | C00.x–C26.x, C30.x–C34.x, C37.x–C41.x, C43.x, C45.x–C58.x, C60.x–C76.x, C81.x–C85.x, C88.x, C90.x–C97.x, | 2 |
| Renal disease | I12.0, I13.1, N03.2-N03.7, N05.2-N05.7, N18.x, N19.x, N25.0, Z49.0-Z49.2, Z94.0, Z99.2 | 2 |
| Moderate or severe liver disease | I85.0, I85.9, I86.4, I98.2, K70.4, K71.1, K72.1, K72.9, K76.5, K76.6, K76.7 | 3 |
| AIDS/HIV | B20.x-B22.x, B24.x | 6 |
| Metastatic solid tumor | C77.x-C80.x | 6 |


**Table 12. Baseline Medications** 

| Class | Drug |
|---|---|
| NSAIDs | Bromfenac, Celecoxib, Diclofenac, Etodolac, Fenoprofen, Flurbiprofen, Ibuprofen, Indomethacin, Ketoprofen, Ketorolac, Naproxen, Meclofenamate, Mefenamic acid, Meloxicam, Nabumetone, Oxaprozin, Piroxicam, Sulindac, Tolmetin |
| Antiplatelets | Aspirin, Clopidogrel, Prasugrel, Ticlopidine, Cilostazol, Abciximab, Tirofiban, Dipyridamole, Ticagrelor |
| PPI | Omeprazole, Pantoprazole, Lansoprazole, Rabeprazole, Esomeprazole, Dexlansoprazole |
| H <sub>2</sub> -receptor antagonists | Cimetidine, Ranitidine, Famotidine, Nizatidine, Roxatidine, Lafutidine |
| Antiarrhythmics | Quinidine, Procainamide, Mexiletine, Propafenone,<br>Flecainide, Amiodarone, Bretylium, Dronedarone,<br>Propranolol, Atenolol, Esmolol, Verapamil, Diltiazem,<br>Sotalol |
| Digoxin | Digoxin |
| Statins | Atorvastatin, Fluvastatin, Lovastatin, Pitavastatin, Pravastatin, Roxuvastatin, Simvastatin |

Table 13. Exclusion Criteria

| Condition | KCD Code or Korean Procedure Codes |
|---|---|
| Valvular AF/ prosthetic | 105, 108, 109, 134, Q23, T820, T826, Z952, Z953, Z954 |
| heart valves | - Korean Procedure Codes: M6580, M6581, M6582, O1791, |
| | O1792, O1793, O1794, O1795, O1796, O1797, O1798, |
| | O1799, M6531, M6532, M6533, O1690, O1730, 1740, |
| | O1750, O1760, O1770, O1781, O1782, O1783, O1810, |
| | O1826 |
| End-stage of chronic | N185, T824, Y602, Y612, Y622, Y841, Z49, Z992, E1022, |
| kidney disease/ dialysis/ | E1122, E1222, E1322, E1422, Z940 |
| kidney transplant | |
| Venous | 1636, 1676, 1801, 1802, 1803, 1808, 1809, 181, 1822, 1823, 1829, |
| thromboembolism | 126 |
| Thyrotoxicosis | E05 |
| Pericarditis | I30, I31, I32 |
| Hypertrophic | I422 |


| Condition | KCD Code or Korean Procedure Codes |
|---|---|
| cardiomyopathy | |
| Hip or knee replacement* | N0711, N0715, N1711, N1715, N1721, N1725, N2070, N2072, N2077, N2710, N2712, N2717, N3710, N3712, N3717, N3720, N3722, N3727, N4710, N4712, N4717, N4720, N4722, N4727 |
| Elective defibrillation/<br>radiofrequency ablation/<br>left atrial appendage<br>occlusion* | M5880, M6540, M6542, M6545, M6547, M6511 |

<sup>[\*</sup>Note] Hip or knee replacement, elective defibrillation, radiofrequency ablation, and left atrial appendage occlusion will be identified using procedure codes.

**Table 14. Blood Transfusion Codes** 

| Condition | Korean procedure code |
|--------------------------------------------|-----------------------|
| Whole Blood | X1001 |
| Whole Blood | X1002 |
| Fresh Liquid Plasma for Whole Blood 320ml | X2011 |
| Fresh Liquid Plasma for Whole Blood 400ml | X2012 |
| Packed RBC for Whole Blood 320ml | X2021 |
| Packed RBC for Whole Blood 400ml | X2022 |
| Washed RBC for Whole Blood 320ml | X2031 |
| Washed RBC for Whole Blood 400ml | X2032 |
| Fresh Frozen Plasma for Whole Blood 320ml | X2041 |
| Fresh Frozen Plasma for Whole Blood 400ml | X2042 |
| Frozen Plasma for Whole Blood 320ml | X2051 |
| Frozen Plasma for Whole Blood 400ml | X2052 |
| Cryoprecipitate for Whole Blood 320ml | X2061 |
| Cryoprecipitate for Whole Blood 400ml | X2062 |
| Platelet rich plasma for whole blood 320ml | X2071 |


Condition Korean procedure code Platelet Rich Plasma for Whole Blood 400ml X2072 Platelet Concentrate for Whole Blood 320ml X2081 Platelet Concentrate for Whole Blood 400ml X2082 Leukocyte Poor Packed RBC for Whole Blood 320ml X2091 Leukocyte Poor Packed RBC for Whole Blood 400ml X2092 Packed WBC for Whole Blood 320ml X2101 Packed WBC for Whole Blood 400ml X2102 Leukocyte Filtered Packed RBC for Whole Blood 320ml X2111 Leukocyte Filtered Packed RBC for Whole Blood 400 ml X2112 Leukocyte Filtered Packed Platelet Concentrate for Whole X2121 Blood 320ml Leukocyte Filtered Packed Platelet Concentrate for Whole X2122 Blood 400ml Red Blood Cells, Cryopreserved and Thawed for Whole blood X2131 320ml Red Blood Cells, Cryopreserved and Thawed for Whole blood X2132 400ml Plasma, Cryoprecipitate Reduced for Whole blood 320ml X2141 X2142 Plasma, Cryoprecipitate Reduced for Whole blood 400ml Fresh Blood X3010

# 9 REFERENCES

1. Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, et al. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015;131(4):e29-322.

- 2. Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation: a major contributor to stroke in the elderly. The Framingham Study. Arch Intern Med. 1987;147(9):1561-4.
- 3. Savelieva I, Bajpai A, Camm AJ. Stroke in atrial fibrillation: update on pathophysiology, new antithrombotic therapies, and evolution of procedures and devices. Ann Med. 2007;39(5):371-91.
- 4. January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC, Jr., et al. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014;64(21):e1-76.
- 5. Hart RG, Pearce LA, Aguilar MI. Meta-analysis: antithrombotic therapy to prevent stroke in patients who have nonvalvular atrial fibrillation. Annals of internal medicine. 2007;146(12):857-67.
- 6. Banerjee A, Marín F, Lip GY. A New Landscape for Stroke Prevention in Atrial Fibrillation. Stroke. 2011:STROKEAHA. 111.617886.
- 7. Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, et al. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl j Med. 2009;2009(361):1139-51.
- 8. Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, et al. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. New England Journal of Medicine. 2011;365(10):883-91.
- 9. Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, et al. Apixaban versus warfarin in patients with atrial fibrillation. New England Journal of Medicine. 2011;365(11):981-92.
- 10. Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, et al. Edoxaban versus warfarin in patients with atrial fibrillation. New England Journal of Medicine. 2013;369(22):2093-104.
- 11. Stürmer T, Wyss R, Glynn RJ, Brookhart MA. Propensity scores for confounder adjustment when assessing the effects of medical interventions using nonexperimental study designs. Journal of internal medicine. 2014;275(6):570-80.
- 12. Austin PC, Stuart EA. Moving towards best practice when using inverse probability of treatment weighting (IPTW) using the propensity score to estimate causal treatment effects in observational studies. Statistics in medicine. 2015;34(28):3661-79.
- 13. Austin PC, Stuart EA. The performance of inverse probability of treatment weighting and full matching on the propensity score in the presence of model misspecification when estimating the effect of treatment on survival outcomes. Statistical methods in medical research. 2017;26(4):1654-70.